CLINICAL TRIAL: NCT06626880
Title: Predictive Value of Scoring System in Neonates with Disseminated Intravascular Coagulation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Bakr Sleem, Resident Doctor of pediatric, Assiut University
Other Study IDs: DIC scoring system in neonates
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Disseminated Intravascular Coagulation; Neonates
MeSH Terms: conditions — Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aims of this study were to investigate underlying diseases associated with neonatal DIC diagnosed on the first 28 days of life, and whether DIC score could predict mortality in neonates.

DETAILED DESCRIPTION:
Disseminated intravascular coagulation (DIC) is a syndrome caused by the activation of blood coagulation, in which systemic intravascular micro thromboses result in multiple organ failure and severe bleeding due to consumption of platelets and coagulation factors [1]. Compared with adults, neonates have an immature coagulation-fibrinolysis system and are prone to complications that cause DIC, such as hypoxia, acidosis, and infection [2]. Additionally, preterm infants have a lower hemostatic profile than term infants, which increases their risk of DIC [3]. However, gold standard interventions and treatments for DIC are lacking in neonatal medicine, Veldman et al. suggested that DIC in neonates is caused by prenatal risk factors such as placental abruption (PA), pregnancy induced hypertension (PIH), and neonatal factors such as sepsis, asphyxia, and interventricular hemorrhage (IVH), along with postnatal factors, such as necrotizing enterocolitis, gastrointestinal perforation, and infection [4]. The Japan Society of Obstetrical, Gynecological & Neonatal Hematology (JSOGNH) revised its diagnostic guidelines for neonatal DIC in 2016 and proposed a DIC scoring system [5]. Anticoagulant therapy, such as antithrombin administration and fresh frozen plasma (FFP), has been used to treat neonatal DIC [6]. Since 2008, recombinant human soluble thrombomodulin (rTM) has emerged as a novel anticoagulant for DIC in Japan [7]. Reversal of the underlying condition is paramount in achieving treatment success in the newborn with DIC. Strategies such as early antibiotic therapy and identification and control of the source of disease in cases of necrotizing enterocolitis, sepsis, and septic shock should always precede interventions directed at normalizing the coagulation system [8]. reports are lacking about diseases associated with neonatal DIC and whether anything predicts mortality in this context. We discuss the clinical andlaboratory criteria using (JSOGNH) scoring system to see if DIC score could predict mortality in neonates.

ELIGIBILITY:
Inclusion Criteria:

1. age at enrollment from the first day of life to 28 days of life.
2. Neonates diagnosed as DIC.

Exclusion Criteria:

1. Neonates born to mothers with ITP.
2. Autoimmune thrombocytopenic patients.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted on neonates diagnosed as DIC based on their clinical and laboratory data. They will be recruited from NICU at Assiut University Children's Hospital from 1/1/2025 to 1/1/2026.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
The aims of this study were to investigate underlying diseases associated with neonatal DIC diagnosed on the first 28 days of life | from 1/1/2025 to 1/1/2026.
whether DIC score could predict mortality in neonates | from 1/1/2025 to 1/1/2026.
  The aims of this study were to investigate underlying diseases associated with neonatal DIC diagnosed on the first 28 days of life, and whether DIC score could predict mortality in neonates.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Hamdy Phd, Professor of hematology, Study Chair — Professor of hematology of Pediatrics Faculty of Medicine - Assiut University; Amira Shalaby Assistant professor, Study Chair — Assistant professor of neonatology Faculty of Medicine - Assiut University

REFERENCES:
- [Background] Veldman A, Fischer D, Nold MF, Wong FY. Disseminated intravascular coagulation in term and preterm neonates. Semin Thromb Hemost. 2010 Jun;36(4):419-28. doi: 10.1055/s-0030-1254050. Epub 2010 Jul 7. PMID 20614393
- [Background] Shirahata A, Mimuro J, Takahashi H, Tsuji H, Kitajima I, Matsushita T, Eguchi Y, Kitamura N, Honda G, Sakata Y. Postmarketing Surveillance of Recombinant Human Soluble Thrombomodulin (Thrombomodulin alpha) in Pediatric Patients With Disseminated Intravascular Coagulation. Clin Appl Thromb Hemost. 2014 Jul;20(5):465-72. doi: 10.1177/1076029614523490. Epub 2014 Feb 20. PMID 24563247
- [Background] Go H, Ohto H, Nollet KE, Kashiwabara N, Ogasawara K, Chishiki M, Hiruta S, Sakuma I, Kawasaki Y, Hosoya M. Risk factors and treatments for disseminated intravascular coagulation in neonates. Ital J Pediatr. 2020 Apr 29;46(1):54. doi: 10.1186/s13052-020-0815-7. PMID 32349778
- [Background] Poralla C, Traut C, Hertfelder HJ, Oldenburg J, Bartmann P, Heep A. The coagulation system of extremely preterm infants: influence of perinatal risk factors on coagulation. J Perinatol. 2012 Nov;32(11):869-73. doi: 10.1038/jp.2011.182. Epub 2011 Dec 8. PMID 22157628
- [Background] Tay SP, Cheong SK, Boo NY. Circulating tissue factor, tissue factor pathway inhibitor and D-dimer in umbilical cord blood of normal term neonates and adult plasma. Blood Coagul Fibrinolysis. 2003 Feb;14(2):125-9. doi: 10.1097/00001721-200302000-00002. PMID 12632021
- [Background] Wada H, Matsumoto T, Yamashita Y. Diagnosis and treatment of disseminated intravascular coagulation (DIC) according to four DIC guidelines. J Intensive Care. 2014 Feb 20;2(1):15. doi: 10.1186/2052-0492-2-15. eCollection 2014. PMID 25520831